CLINICAL TRIAL: NCT01053039
Title: The Use of Intrathecal Morphine in the Management of Acute Pain Following Decompressive Lumbar Spinal Surgery: A Randomized Controlled Trial
Brief Title: The Use of Intrathecal Morphine in the Management of Acute Pain Following Decompressive Lumbar Spinal Surgery
Acronym: ITMP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Stephan du Plessis, Clinical Assistant Professor, Department of Clinical Neurosciences, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22518
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Acute Pain Following Decompressive Lumbar Spinal Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrathecal Morphine (Active Comparator): Treatment group to receive 0.2mg of intrathecal morphine followed by PCA morphine.
  Interventions: Drug: Intrathecal Morphine
- Intrathecal Saline (Placebo Comparator): The control group will receive intrathecal saline followed by PCA. All patients will receive a standardized postoperative regimen.
  Interventions: Drug: Intrathecal Saline

INTERVENTIONS:
Drug: Intrathecal Morphine — Treatment group to receive 0.2mg of intrathecal morphine followed by PCA morphine.
  Other Names: Epimorph
  Arms: Intrathecal Morphine
Drug: Intrathecal Saline — The control group will receive intrathecal saline followed by PCA. All patients will receive a standardized postoperative regimen.
  Arms: Intrathecal Saline

SUMMARY:
The primary aim of this study is to assess the impact of intrathecal morphine on post-operative pain following instrumented fusion for degenerative lumbar spine disease. Secondary objectives of this study aim to assess side effects, overall narcotic use and duration of hospital stay following administration of intrathecal morphine.

Based on our literature review, we expect a significant improvement in pain scores and functional status and minimal side effects with the use of intrathecal morphine. With improved pain and function we would also expect shorter hospital stays in those patients receiving intrathecal morphine.

DETAILED DESCRIPTION:
Adult patients (>18 yrs or older) undergoing instrumented fusion for degenerative lumbar spine disease will be recruited and randomized to receive one of two treatments. The first group will receive an injection of morphine (200mcg) into the intrathecal space at the time of the operation. The second group will receive a saline injection. The pharmacy will prepare the aforementioned injections and deliver them to the operating room to ensure all parties are blinded. Both groups will then have a standardized analgesic regimen (including PCA morphine and parenteral analgesics) available to them in the post-operative period. Each group will be followed at regular intervals post-operatively. At each follow-up, visual analogue pain scores, side effects and narcotic use will be assessed. Patients will also have a daily functional assessment which will dictate the time of discharge. Hospital stay will be measured from time of admission to time where patient no longer requires acute hospital care based on the functional assessment.

ELIGIBILITY:
Inclusion Criteria:

* age 18yrs or older
* elective surgery for instrumented fusion of the lumbar spine for stenosis (< 5 levels)
* with back and/or leg pain
* patients who meet ASA class 1 or 2

Exclusion Criteria:

* Patients unable to speak english
* known allergies to morphine or other opioids
* spinal surgery other than lumbar spine surgery
* history of severe respiratory illness including COPD and asthma
* history of obstructive sleep apnea
* pregnancy
* lumbar procedures performed in minimally invasive fashion
* patients lacking mental capacity to use PCA
* patients on sustained release narcotics
* patients undergoing revision of previous instrumented lumbar spine surgery
* patients with psychiatric disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-01; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The primary aim of this study is to assess the impact of intrathecal morphine on post-operative pain following instrumented fusion for lumbar spinal stenosis. | Pre-op to discharge

SECONDARY OUTCOMES:
Secondary objectives of this study aim to assess side effects, overall narcotic use and duration of hospital stay following administration of intrathecal morphine. | Pre-op to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Stephan J du Plessis, MD, FRCSC, Principal Investigator — Chairman, University of Calgary Spine Program
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada